CLINICAL TRIAL: NCT07250230
Title: Effect of Perioperative High-dose Transdermal Nicotine Patch on Pain Sensitivity Among Male Abstinent Tobacco Smokers Undergoing Thoracic Surgery: A Randomized Controlled Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: meinihaokan
Record Dates: First submitted 2025-06-07; First posted 2025-11-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-06

CONDITIONS: Nicotine Dependence; Thoracic Diseases; Analgesia
MeSH Terms: conditions — Tobacco Use Disorder; Thoracic Diseases; Agnosia | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotine patch group (group N) (Experimental): Based on analgesia in the control group, the patients were given a nicotine patch every day, 24 hours before surgery and 48 hours after surgery, placed on the patient's arm, chest, or back, and the skin was cleaned before the patch. Different doses of nicotine patches are given depending on the number of cigarettes smoked by the patient (one 21 mg patch for every 20 cigarettes, 42 mg patch for patients who smoke ≥ 40 cigarettes per day)
  Interventions: Drug: Nicotine patch
- Control group (Group C) (No Intervention): On the basis of conventional analgesia, patients were given a placebo patch without any drug effect every day 24 hours before surgery and 48 hours after surgery, and the shape, weight, and position of the patch were consistent with those of the experimental group

INTERVENTIONS:
Drug: Nicotine patch — Based on analgesia in the control group, the patients were given a nicotine patch every day, 24 hours before surgery and 48 hours after surgery, placed on the patient's arm, chest, or back, and the skin was cleaned before the patch. Different doses of nicotine patches are given depending on the number of cigarettes smoked by the patient (one 21 mg patch for every 20 cigarettes, 42 mg patch for patients who smoke ≥ 40 cigarettes per day)
  Arms: Nicotine patch group (group N)

SUMMARY:
Globally, approximately 230 million adults undergo surgical procedures each year, with around 30% of patients maintaining smoking habits prior to surgery. Extensive clinical research has confirmed that tobacco exposure is a significant independent risk factor for perioperative complications. Epidemiological data indicate that long-term smokers experience a significantly higher all-cause mortality rate during hospitalization, approximately 20% greater than non-smokers, while the incidence of postoperative complications is 40% higher. Consequently, international guidelines universally recommend the establishment of standardized preoperative smoking cessation programs for surgical patients. Nicotine withdrawal, a typical clinical manifestation during smoking cessation, involves symptoms across multiple systems: neuropsychiatric symptoms such as mood depression, sleep disturbances, and irritability; autonomic dysfunction leading to postural dizziness and bradycardia; and metabolic dysregulation resulting in increased appetite and weight gain. Notably, these withdrawal symptoms exhibit a significant time-dependent pattern, typically peaking 24-72 hours after cessation. Multicenter studies have demonstrated that tobacco-dependent patients experience an average increase of IV Abstract 35-45% in opioid consumption within 24 hours postoperatively, with the duration of analgesic requirements extended by approximately 25%. However, some patients suffer from severe adverse reactions to opioids (e.g., nausea, vomiting, confusion), making the use of adjuvant medications for multimodal analgesia and optimized pain management particularly crucial. By the late 20th century, the analgesic properties of nicotine, a primary component of tobacco, were systematically studied and applied in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male, aged 18-75 years, with a body mass index (BMI) of 18-28 kg/m2 Between;
2. Thoracoscopic lobectomy/segmental/wedge resection under general anesthesia;
3. American Society of Anesthesiologists (ASA) classifications I-III Level;
4. Regular smoking for more than 2 years, smoking more than 10 cigarettes per day in the past 6 months, and not successfully quitting smoking within 1 month (after admission, the doctor and nurse informed the smoking cessation plan to intervene before starting to stop smoking or 1 ≤ cigarette count ≤ 10 cigarettes/day in the past month), FTND score ≥ 2;
5. No severe respiratory diseases, no serious cardiovascular and cerebrovascular diseases (hypertension is treated with SBP ≤ 160mmHg, DBP ≤ 90mmHg after systemic treatment);
6. Obtain informed consent.

Exclusion Criteria:

1. Those who have a history of alcoholism, long-term use of sedatives or analgesics;
2. Patients with psychiatric and nervous system diseases (such as Parkinson's, depression, schizophrenia) and severe audio-visual dysfunction before surgery;
3. Preoperative systolic blood pressure > 180mmHg or diastolic blood pressure > 110mmHg;
4. Patients who were converted to thoracotomy during thoracoscopic surgery
5. Patients who are transferred to the intensive care unit after surgery;
6. Patients who refuse to use analgesic pump treatment/do not configure the analgesic pump according to regulations;
7. Patients who have self-removed patches/short hospital stay resulting in a postoperative observation time of < 48 hours

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Analgesic pump dosage in (ml) for Postoperative pain | 48 hours
  Analgesic pump dosage at 1, 6, 24, 48 hours postoperative operation (ml)

CONTACTS AND LOCATIONS:
Overall Officials: Jiaqiang Zhang, PHD, Study Chair — Henan Provincial People's Hospital
Locations (1):
- Department of Anaesthesiology and Perioperative Medicine, People's Hospital of Zhengzhou University, Henan Provincial People's Hospital, Zhengzhou, Henan, Zhengzhou, Henan, China